CLINICAL TRIAL: NCT03457467
Title: Clinical Study of Apatinib Mesylate Combined With Stereotactic Body Radiation Therapy in the Treatment of Oligometastasis of Breast Cancer
Brief Title: Clinical Study of Apatinib Combined With SBRT Therapy in the Treatment of Oligometastasis of Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yan Li (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yan Li, assistant director physician, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-BC-20170323
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: oligometacosis; anti-angiogenic; apatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+apatinib group (Experimental): Apatinib mesylate tablets: 500mg / day, 28 days / cycle, follow-up to the progress of the disease, toxicity intolerable or patients require withdrawal; SBRT: according to the different treatment sites given the corresponding dose: 1200cGy × 4 times or 800cGy × 7 times, or according to the specific situation dose adjustment.
  Interventions: Drug: Apatinib; Radiation: SBRT

INTERVENTIONS:
Drug: Apatinib — Apatinib 500 mg is administered orally daily, until disease progression or untolerable toxicity
  Other Names: Apatinib Mesylate Tablets
Radiation: SBRT — according to the different treatment sites given the corresponding dose: 1200cGy × 4 times or 800cGy × 7 times, or according to the specific situation dose adjustment
  Other Names: Stereotactic body radiotherapy

SUMMARY:
The treatment of the patients with metastatic breast cancer remains a major problem. However, there is an intermediate state between the primary tumor and distant metastases called oligometastasis. Current research indicates that good local control of oligometastasis can be obtained with Stereotactic body radiotherapy (SBRT) Can not prolong the long-term survival of patients. Researchers believe that after SBRT treatment of patients with oligometacosis in breast cancer, it is necessary to explore whether the anti-angiogenic therapy targeted drug apatinib can reduce the occurrence of new lesions and prolong the survival of patients.

DETAILED DESCRIPTION:
The treatment of the patients with metastatic breast cancer remains a major problem. However, there is an intermediate state between the primary tumor and distant metastases called oligometastasis. Current research indicates that good local control of oligometastasis can be obtained with Stereotactic body radiotherapy (SBRT) Can not prolong the long-term survival of patients. Researchers believe that after SBRT treatment of patients with oligometacosis in breast cancer. So, through the detection of microRNA in the primary lesion of breast cancer patients with oligometastasis to screen the patients with oligomerization and potential multiple metastases; explore the existing medical treatment, based on the control of local lesions by SBRT, the use of apatinib anti-angiogenic targeted maintenance therapy, with a view to reducing the incidence of new lesions, thereby prolonging the patient's survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old women; 2. Histologically confirmed breast cancer; 3 weeks before enrollment ECOG PS score: 0-2 points; 4. systemic metastasis lesions ≤ 5, Stereotactic body radiotherapy before receiving medical treatment to achieve partial relief or stable disease; 5. Appropriate hematological parameters and liver and kidney function: absolute neutrophil ≧ 1.5 × 109 / L; platelet count ≧ 75 × 109 / L; serum total bilirubin ≦ 1.5 × upper limit of normal; AST and ALT ≦ 2.5 × upper limit of normal (if liver dysfunction) 6. Subject voluntarily joined the study and signed the informed consent form.

Exclusion Criteria:

1. After the above image examination of the whole body metastasis lesions ≥ 6;
2. Have received one or more palliative chemotherapy regulators failed;
3. Patients with a high risk of bleeding: active gastric digestive ulcer in the stomach with fecal occult blood (++); those with a history of melena and / or vomiting within 3 months; persons with abnormal coagulation and bleeding tendency; 3-4 grade hypertension patients;

5. Renal insufficiency 3 and above patients; 6. Hand-foot syndrome ≥ 3 or more patients; 7. There are uncontrolled concomitant diseases in the first 6 months of the study, including unstable angina pectoris, acute myocardial infarction, cerebrovascular accident and so on; 8. Pregnant or breastfeeding patients, or who have fertility without taking contraceptive measures; 9. A history of malignancy, but disease-free survival of more than 5 years; 10. Concurrent with other anti-cancer therapies or other interventional clinical trials; 11. Patients unable to follow the study due to psychological, family-living social reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer
Enrollment: 30 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Approximately 3 year
  OS is defined as the length of time from random assignment to death or to last contact.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Approximately 2 year
  time from randomization to documented progressive disease or death due to any cause, whichever occurs first
Adverse Events(AEs) | Approximately 2 years
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hellman S. Karnofsky Memorial Lecture. Natural history of small breast cancers. J Clin Oncol. 1994 Oct;12(10):2229-34. doi: 10.1200/JCO.1994.12.10.2229. No abstract available. PMID 7931493
- [Background] Milano MT, Zhang H, Metcalfe SK, Muhs AG, Okunieff P. Oligometastatic breast cancer treated with curative-intent stereotactic body radiation therapy. Breast Cancer Res Treat. 2009 Jun;115(3):601-8. doi: 10.1007/s10549-008-0157-4. Epub 2008 Aug 22. PMID 18719992
- [Background] Lo SS, Fakiris AJ, Chang EL, Mayr NA, Wang JZ, Papiez L, Teh BS, McGarry RC, Cardenes HR, Timmerman RD. Stereotactic body radiation therapy: a novel treatment modality. Nat Rev Clin Oncol. 2010 Jan;7(1):44-54. doi: 10.1038/nrclinonc.2009.188. Epub 2009 Dec 8. PMID 19997074
- [Background] Lo SS, Fakiris AJ, Teh BS, Cardenes HR, Henderson MA, Forquer JA, Papiez L, McGarry RC, Wang JZ, Li K, Mayr NA, Timmerman RD. Stereotactic body radiation therapy for oligometastases. Expert Rev Anticancer Ther. 2009 May;9(5):621-35. doi: 10.1586/era.09.15. PMID 19445579
- [Background] Lussier YA, Xing HR, Salama JK, Khodarev NN, Huang Y, Zhang Q, Khan SA, Yang X, Hasselle MD, Darga TE, Malik R, Fan H, Perakis S, Filippo M, Corbin K, Lee Y, Posner MC, Chmura SJ, Hellman S, Weichselbaum RR. MicroRNA expression characterizes oligometastasis(es). PLoS One. 2011;6(12):e28650. doi: 10.1371/journal.pone.0028650. Epub 2011 Dec 13. PMID 22174856
- [Background] Elson-Schwab I, Lorentzen A, Marshall CJ. MicroRNA-200 family members differentially regulate morphological plasticity and mode of melanoma cell invasion. PLoS One. 2010 Oct 4;5(10):e13176. doi: 10.1371/journal.pone.0013176. PMID 20957176
- [Background] Dykxhoorn DM, Wu Y, Xie H, Yu F, Lal A, Petrocca F, Martinvalet D, Song E, Lim B, Lieberman J. miR-200 enhances mouse breast cancer cell colonization to form distant metastases. PLoS One. 2009 Sep 29;4(9):e7181. doi: 10.1371/journal.pone.0007181. PMID 19787069
- [Background] Wong AC, Watson SP, Pitroda SP, Son CH, Das LC, Stack ME, Uppal A, Oshima G, Khodarev NN, Salama JK, Weichselbaum RR, Chmura SJ. Clinical and molecular markers of long-term survival after oligometastasis-directed stereotactic body radiotherapy (SBRT). Cancer. 2016 Jul 15;122(14):2242-50. doi: 10.1002/cncr.30058. Epub 2016 May 20. PMID 27206146